CLINICAL TRIAL: NCT02983812
Title: Developing Enhanced Prediction Models to Identify Patients at Risk for Hospital Readmission by Collecting Patient-Generated Health Data
Brief Title: Developing Enhanced Prediction Models
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 825189
Record Dates: First submitted 2016-11-16; First posted 2016-12-06 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infraction or Chest Pain; Chronic Obstructive Pulmonary Disease (COPD); Congestive Heart Failure (CHF); Diabetes; Pneumonia
MeSH Terms: conditions — Chest Pain; Pulmonary Disease, Chronic Obstructive; Heart Failure; Diabetes Mellitus; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Activity Monitoring - Smartphone: Patients in the activity monitoring - smartphone group will be randomly assigned to track their data using a smartphone app (which collects step counts) for 6 months. There will be no intervention for either group, both are being passively monitored.
- Activity Monitoring - Wearable: Patients in the activity monitoring - wearable device group will be randomly assigned to track their data using a wearable activity tracker (which collects step counts and sleep patterns/duration). There will be no intervention for either group, both are being passively monitored.

SUMMARY:
In this study, patients will be prospectively enrolled for data collection to design prediction models that integrate claims data (inpatient, outpatient, and pharmacy), electronic health record data (on clinical, social, and behavioral indicators), and patient-generated activity data. Patients will be randomized to use either a smartphone or a wearable activity tracking device to capture patient-generated health data.

DETAILED DESCRIPTION:
Many hospital readmissions could be prevented if higher risk patients were identified and effective interventions then targeted towards these individuals. However, most existing claims-based predictive models perform poorly and do not provide timely and actionable information. In this study, researchers will prospectively enroll patients for data collection to design prediction models that integrate claims data (inpatient, outpatient, and pharmacy), electronic health record data (on clinical, social, and behavioral indicators), and use wearable devices or smartphones to collect patient-generated data (physical activity and sleep patterns). Patients will be randomized to use either a smartphone or a wearable activity tracking device to capture patient-generated health data.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older
2. Be able to provide informed consent
3. Be admitted to the Hospital of the University of Pennsylvania or Penn Presbyterian Medical Center
4. Have a smartphone or tablet compatible with activity tracking devices
5. Plan to be discharged to home

Exclusion Criteria:

Have no medical condition which prohibits them from ambulating or plan for any medical procedure over the next 6 months that would prohibit them from ambulating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from adults admitted to one of the University of Pennsylvania Health System hospitals. Patients will be invited to participate by a member of the research team prior to hospital discharge.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Hospital readmission within 30 days of discharge | 30 days
  Patient readmission within 30 days of initial discharge

SECONDARY OUTCOMES:
The secondary outcome measures include re-hospitalization within 90 days of discharge. | 90 days
  Patient readmission within 90 days of initial discharge
Re-hospitalization within 6 months of discharge | 6 months
  Patient readmission within 6 months of initial discharge
Emergency department visits within 6 months of discharge | 6 months
  Patient visit to the emergency department within 6 months of initial discharge
Total health care cost utilization in 6 months after discharge | 6 months
  The cost of health care services for patient within 6 months of initial discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Derived] Patel MS, Polsky D, Kennedy EH, Small DS, Evans CN, Rareshide CAL, Volpp KG. Smartphones vs Wearable Devices for Remotely Monitoring Physical Activity After Hospital Discharge: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Feb 5;3(2):e1920677. doi: 10.1001/jamanetworkopen.2019.20677. PMID 32031643
- [Derived] Evans CN, Volpp KG, Polsky D, Small DS, Kennedy EH, Karpink K, Djaraher R, Mansi N, Rareshide CAL, Patel MS. Prediction using a randomized evaluation of data collection integrated through connected technologies (PREDICT): Design and rationale of a randomized trial of patients discharged from the hospital to home. Contemp Clin Trials. 2019 Aug;83:53-56. doi: 10.1016/j.cct.2019.06.018. Epub 2019 Jun 29. PMID 31265915